CLINICAL TRIAL: NCT06144086
Title: A Multi-center, Single-arm, Open-label Phase 2 Trial of Foscenvivint in Liver Cirrhosis Patients Caused by HIV/HCV Co-infection with Hemophilia
Brief Title: A Phase 2 Trial of Foscenvivint in Liver Cirrhosis Patients Caused by HIV/HCV Co-infection with Hemophilia (OP-724-H201)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kiminori Kimura, MD (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor-Investigator, Kiminori Kimura, MD, Director, Department of Hepatology, Komagome Hospital
Organization: Komagome Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-724-H201; jRCT2031230461 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Hemophilia; HIV/HCV co-infection
MeSH Terms: conditions — Liver Cirrhosis; Hemophilia A | interventions — ICG 001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Foscenvivint (Experimental): Foscenvivint 280 mg/m2, twice a week for 24 weeks
  Interventions: Drug: Foscenvivint

INTERVENTIONS:
Drug: Foscenvivint — Administered by intravenous (IV) infusion over 3-4 hours
  Other Names: CBP-beta-catenin inhibitor; OP-724; PRI-724 (former name)

SUMMARY:
This is a phase 2 trial of foscenvivint in liver cirrhosis patients caused by HIV/HCV co-infection with hemophilia to evaluate the efficacy, safety and pharmacokinetics.

DETAILED DESCRIPTION:
This is designed a multi-center, single-arm, open-label trial of foscenvivint administered intravenously twice a week for 24 weeks. A follow up visit will be conducted 4 weeks after the last administration.

Liver cirrhosis patients due to co-infection of HIV and HCV with hemophilia who have a Child-Pugh classification of A or B are included.

ELIGIBILITY:
Key Inclusion Criteria

* Hemophilia patients with liver cirrhosis caused by HIV/HCV co-infection that fall under the following 1) and 2):

  1. Serum HIV-RNA positive or HIV antibody positive patients (maintaining HIV-RNA < 200 copies/mL and CD4 positive T lymphocyte count >= 200 cells/µL at screening).
  2. Regarding HCV, patients who had passed >= 12 months after achieving SVR at registration.
* Patients with Child-Pugh classification A or B (Child-Pugh score 5-9).
* Patients who meet at least one of 1) to 2) for diagnosis of liver cirrhosis:

  1. Liver stiffness measurement by FibroScan is >= 12.5 kPa (Fibrosis stage F4) at screening.
  2. Abdominal CT scan shows changes in liver shape and/or portal hypertension.
* Patients with Performance Status 0-2.

Key Exclusion Criteria

* Patients with liver cirrhosis of which cause is not HCV or unknown.
* Patients with esophageal gastric varices judged to require treatment by endoscopic examinations at screening.
* Patients with complication or history of malignant tumor (within 3 years before registration).
* Patients who have undergone liver transplantation or other organ transplantation (including bone marrow transplantation).
* Patients with active AIDS-indicator disease that require treatment.

Ages: 18 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
ALBI score | Baseline to 24 weeks after administration
  Change from baseline in ALBI score at 24 weeks after administration.
  ALBI score = (log10 bilirubin [mg/dL] x 17.1) x 0.66 + (albumin [g/dL] x 10 x -0.085)

SECONDARY OUTCOMES:
Child-Pugh score | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in Child-Pugh score at 12, 24 and 28 weeks after administration.
  Child-Pugh score is determined by scoring the following five clinical measures.
  Encephalopathy: None = 1 point, Grade 1 and 2 = 2 points, Grade 3 and 4 = 3 points
  Ascites: None = 1 point, slight = 2 points, moderate = 3 points
  Bilirubin: < 2 mg/dL = 1 point, 2 to 3 mg/dL = 2 points, > 3 mg/dL = 3 points
  Albumin: > 3.5 g/dL = 1 point, 2.8 to 3.5 g/dL = 2 points, < 2.8 g/dL = 3 points
  Prothrombin Time (%): > 70% = 1 point, 40 to 70% = 2 points, < 40% = 3 points
ALBI score | Baseline to 12 and 28 weeks after administration
  Change from baseline in ALBI score at 12 and 28 weeks after administration.
Liver stiffness measurement by FibroScan | Baseline to 12 and 24 weeks after administration
  Change from baseline in Liver stiffness measurement by FibroScan at 12 and 24 weeks after administration.
Serum fibrosis markers | Baseline to 12 and 24 weeks after administration
  Change from baseline in Serum fibrosis markers at 12 and 24 weeks after administration.
Serum albumin | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in serum albumin at 12, 24 and 28 weeks after administration.
Serum bilirubin | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in serum bilirubin at 12, 24 and 28 weeks after administration.
PT% | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in PT% at 12, 24 and 28 weeks after administration.
MELD score | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in MELD score at 12, 24 and 28 weeks after administration.
  The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. The higher the score, the more serious the subject's disease. MELD is calculated according to the following formula:
  MELD score = 3.78 x ln(serum bilirubin [mg/dL]) + 11.2 x ln(PT-INR) + 9.57 x ln(serum creatinine [mg/dL]) + 6.43
FIB-4 index | Baseline to 12, 24 and 28 weeks after administration
  Change from baseline in FIB-4 index at 12, 24 and 28 weeks after administration.
  FIB-4 index = (Age [years] x AST [U/L]) / (Platelet Count [10*9/L] x √ ALT [U/L] )
mALBI grade | Baseline to 12, 24 and 28 weeks after administration
  Percentage of subjects who achieved >= 1 stage improvement in mALBI grade from baseline at 12, 24 and 28 weeks after administration.
  Based on ALBI score, mALBI grade is classified into Grade 1 to 3 shown below.
  mALBI grade: Grade 1: <=-2.60; Grade 2a: >-2.60 to <-2.27; Grade 2b: >=-2.27 to -1.39; Grade 3: >-1.39
Achievement in Child-Pugh classification | Baseline to 12, 24 and 28 weeks after administration
  Percentage of subjects who changed from grade B at baseline to grade A at 12, 24 and 28 weeks after administration in Child-Pugh classification.
  Based on the total points in Child-Pugh score (scale range 5-15 points, the severity increases sequentially from 5 to 15 points), the severity of the disease is classified into Grade A to C shown below.
  Child-Pugh classification:
  Grade A: 5 to 6 points -> Compensated cirrhosis; Grade B: 7 to 9 points -> Decompensated cirrhosis; Grade C: 10 to 15 points -> Decompensated cirrhosis
Achievement in Child-Pugh score | Baseline to 12, 24 and 28 weeks after administration
  Percentage of subjects who achieved >= 2 points improvement from baseline in Child-Pugh score at 12, 24 and 28 weeks after administration.
Achievement in Child-Pugh classification and score | Baseline to 12, 24 and 28 weeks after administration
  Percentage of subjects who changed from grade B to grade A in Child-Pugh classification and achieved >= 2 points improvement in Child-Pugh score from baseline at 12, 24 and 28 weeks after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Kiminori Kimura, MD, Principal Investigator — Tokyo Metropolitan Komagome Hospital
Locations (3):
- Japan (3):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No